CLINICAL TRIAL: NCT05678647
Title: Randomized Open Comparative Trial of Oral Sucrosomial Iron (SiderAl Forte®) and Oral Iron Sulphate (Duroferon®) to Blood Donors.
Brief Title: Sucrosomial Iron and Iron Sulphate to Blood Donors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Karin Schneider, MD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOU2022-00167 980506
Record Dates: First submitted 2022-11-30; First posted 2023-01-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Blood Donation
MeSH Terms: interventions — sucrosomial iron; Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: Drugs:
  Oral sucrosomial Iron (SiderAl Forte®) and oral iron sulphate (Duroferon®) to blood donors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral sucrosomial Iron (SiderAl Forte®) (Experimental): Oral sucrosomial Iron (SiderAl Forte®) is given to blood donors after blood donation
  Interventions: Drug: Sucrosomial Iron
- Oral iron sulphate (Duroferon®) (Active Comparator): Oral iron sulphate (Duroferon®) is given to blood donors after blood donation
  Interventions: Drug: Iron Sulfate

INTERVENTIONS:
Drug: Sucrosomial Iron — 20 capsules of Sucrosomial Iron 30 mg is given after blood donation
  Other Names: SiderAl Forte®
  Arms: Oral sucrosomial Iron (SiderAl Forte®)
Drug: Iron Sulfate — 20 tablets of oral iron sulphate (Duroferon®) 100 mg is given after blood donation
  Other Names: Duroferon®
  Arms: Oral iron sulphate (Duroferon®)

SUMMARY:
2 different oral iron supplementations after blood donation are compared.

DETAILED DESCRIPTION:
Iron depletion is common in regular blood donors. During a blood donation the donor loses 200-250 mg iron. The routine at our donor sites is to give donors 20 tablets of iron sulphate (Duroferon®) 100 mg after blood donation.

In this study we will compare two different iron supplementations given after blood donation. 60 donors are given oral sucrosomial Iron (SiderAl Forte®) and 60 donors are given oral iron sulphate (Duroferon®) after 4 successive blood donation.

The primary purpose of this study is to compare the side effects of sucrosomial Iron and iron sulphate and to investigate if the iron balance can be maintained with sucrosomial iron.

After each blood donation the donors are asked to answer a questionary with questions about side effects and symptoms of Restless legs syndrome/Willis-Ekbom (symptoms associated with iron deficiency).

ELIGIBILITY:
Inclusion Criteria:

Blood donors at Uppsala University hospital wo have been donating blood regularly the last two years are eligible to participate in the study.

Exclusion Criteria:

Donors who cannot be accepted for blood donation anymore because they do not fulfill the Swedish criteria for blood donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Side effects | One year
  The side effects are compared. At every visit the donors are asked to answer a questionary with questions about side effects.
  The amount and severity of the side effects will be compared between the two groups with different iron supplementations.

SECONDARY OUTCOMES:
Symptoms | One year
  Symptoms of Restless legs syndrome/Willis-Ekbom syndrom. At every visit the donors are asked to answer a questionary with questions about symptoms of restless legs.
  The amount and severity of the symptoms of the two groups with different iron supplementations will be compared.
Iron balance | One Year
  Laboratory analyzes

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Lubenow, PhD, Principal Investigator — Clinical Immunology and Transfusion Medicine Uppsala University Hospital
Locations (1):
- Clinical Immunology and Transfusion Medicine, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared.

REFERENCES:
- [Background] Gomez-Ramirez S, Brilli E, Tarantino G, Munoz M. Sucrosomial(R) Iron: A New Generation Iron for Improving Oral Supplementation. Pharmaceuticals (Basel). 2018 Oct 4;11(4):97. doi: 10.3390/ph11040097. PMID 30287781
- [Background] Fabiano A, Brilli E, Mattii L, Testai L, Moscato S, Citi V, Tarantino G, Zambito Y. Ex Vivo and in Vivo Study of Sucrosomial(R) Iron Intestinal Absorption and Bioavailability. Int J Mol Sci. 2018 Sep 12;19(9):2722. doi: 10.3390/ijms19092722. PMID 30213039
- [Background] Birgegard G, Schneider K, Ulfberg J. High incidence of iron depletion and restless leg syndrome (RLS) in regular blood donors: intravenous iron sucrose substitution more effective than oral iron. Vox Sang. 2010 Nov;99(4):354-61. doi: 10.1111/j.1423-0410.2010.01368.x. PMID 20598107
- [Background] Pisani A, Riccio E, Sabbatini M, Andreucci M, Del Rio A, Visciano B. Effect of oral liposomal iron versus intravenous iron for treatment of iron deficiency anaemia in CKD patients: a randomized trial. Nephrol Dial Transplant. 2015 Apr;30(4):645-52. doi: 10.1093/ndt/gfu357. Epub 2014 Nov 13. PMID 25395392
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159